CLINICAL TRIAL: NCT06050655
Title: The Efficacy of Lingual Aligners in Adults: a Pilot Study.
Brief Title: The Efficacy of Lingual Aligners in Adults.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Fabiana Mutzenberg, Principal investigator, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-D0045
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Malocclusion, Angle Class I
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with Angle Class I malocclusion (Experimental): * Adults older than 18 years old
  * About to undergo orthodontic treatment
  Interventions: Device: Lingual aligners

INTERVENTIONS:
Device: Lingual aligners — orthodontic treatment with lingual aligners

SUMMARY:
The goal of this clinical trial is to test the effectiveness of lingual aligners in adults.

The main question to answer is:

- Are lingual aligners effective in achieving desired and predicted tooth movements?

DETAILED DESCRIPTION:
The aim of this pilot study is to assess the effectiveness and the accuracy of lingual aligners by evaluating the discrepancy between the predicted and the achieved amounts of tooth movements.

Also:

* Patient discomfort and pain
* Appliance defects
* Patient compliance
* Chair and treatment time

Key inclusion criteria:

* Adults older than 18 years old
* About to undergo orthodontic treatment

Key exclusion criteria:

* Patients with tooth extractions or tooth agenesis with space closure
* Patients with surface enamel defects
* Pregnant patients
* Syndromic patients or those with cleft lip and/or palate
* Patients with metabolic diseases

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years old
* About to undergo orthodontic treatment

Exclusion Criteria:

* Patients with tooth extractions or tooth agenesis with space closure
* Patients with surface enamel defects
* Pregnant patients
* Syndromic patients or those with cleft lip and/or palate
* Patients with metabolic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Tooth movement | At the end of study completion, an average of 10 months.
  Tooth movement in the three planes of space measured millimetrically and with degrees, depending on the type of tooth movement

SECONDARY OUTCOMES:
Patient discomfort / pain | Each patient visit, through study completion, an average of 10 months
  Rate of Patient discomfort using the visual assessment scale
Appliance defects | Each patient visit, through study completion, an average of 10 months
  Rate of Breakage or cracking of the aligners
Patient compliance | Each patient visit, through study completion, an average of 10 months
  Indice of Patient compliance evaluated with a questionnaire
Chair and treatment time | Each patient visit, through study completion, an average of 10 months .
  The amount of time the patient spends on the dental chair at each visit measured in minutes; and treatment length in months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
Primary participant data will only be shared with other researchers upon reasonable request